CLINICAL TRIAL: NCT00829491
Title: Denver Health Cardiovascular Prevention Program
Brief Title: Denver Health Cardiovascular Disease (CVD) Prevention Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Denver Health and Hospital Authority (Other)
Collaborators: Colorado Department of Public Health and Environment (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 07-0020
Record Dates: First submitted 2009-01-23; First posted 2009-01-27 (Estimated); Last update posted 2012-07-17 (Estimated); Status verified 2012-07

CONDITIONS: Cardiovascular Disease
Keywords: Cardiovascular Disease Prevention; Behavior change; Risk Reduction
MeSH Terms: conditions — Cardiovascular Diseases; Risk Reduction Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: CVD risk reduction program — Participants will be selected through review of the DH administrative databases or by referral from their primary care provider. After completion of the forms, the navigator and client will discuss potential CVD risk reduction activities and programs available through this program for the client to participate in. Potential activities will include self-monitoring using self-help tools,healthy nutrition and exercise activities, community-based exercise programs using the recreation centers in the community, and referral to the Colorado Quitline for smoking cessation activities. Follow-up questionnaires will be completed at 6 and 12 months after enrollment to assess changes in levels of exercise, dietary patterns, and beliefs and attitudes about behavioral change.
  Other Names: CDPHE, CCPD grants programs.

SUMMARY:
The objective of the Denver Health CVD Prevention Program is to assess the effectiveness of developing an enhanced cardiovascular disease prevention program in a community health care setting.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the leading cause of mortality in Colorado.[1] This is especially true in the Latino population who are at greater risk for CVD compared to non-Latino whites, and suffer more premature CVD deaths.[2] Among persons less than 34 years, Latinos are four times more likely to die from heart disease than non-Latino whites, a disparity that lessens but does not disappear with age (1.5 ratios among persons 55 - 64 yrs old). Recently, the INTERHEART study demonstrated that 90% of the population attributable risk is due to established modifiable risk factors (smoking, dyslipidemia, hypertension, diabetes, obesity, psychosocial factors, daily consumption of fruits and vegetables, regular alcohol consumption and regular physical activity).[3] Many individuals in the general population have one or more risk factors for CVD and over 90% of CVD events occur in individuals with at least one risk factor,[3, 4] with few events occurring in individuals with no risk factors, thus supporting the notion of focusing prevention activities on individuals at higher risk for CVD.

Reducing the risk of CVD is part of Colorado's strategic plan. Programs are needed that offer provide enhanced patient-centered CVD prevention services using paraprofessionals and thus assisting health care providers (i.e., physicians, midlevels) in addressing preventive health care issues. Early identification of CVD risk is paramount in order to reach those who need the appropriate treatment. In this regard, NCEP guidelines recommend the utilization of the Framingham Risk Score (FRS) as the basis to identify patients with an increased 10-year risk for CVD events.

Despite evidence of the effectiveness of preventive services and the development of published national guidelines,[5, 6] rates of delivery of preventive services remain low.[7] The most common barriers identified are the lack of time during the office visit, inadequate insurance reimbursement, patient refusal to discuss or comply with recommendations, and lack of physician expertise in counseling techniques.[8-12] At Denver Community Health Services (DCHS), a department of Denver Health (DH), an additional barrier includes socioeconomic issues associated with a low-income population with ethnically diverse issues. Thus, delivering CVD preventive services often takes a lower priority during an office visit in a busy clinical practice. However, proactively identifying individuals at risk of CVD and involving them in their own care should increase awareness of CVD risk factors and as such assist in reducing the burden of CVD in the community.

Denver Public Health (DPH) in collaboration with DCHS will implement a comprehensive cardiovascular risk assessment and prevention treatment plan among three westside community health centers. In order to improve CVD risk reduction, this demonstration project will a) develop a CVD registry to be able to identify at risk individuals, b) engage high-risk patients to participate in CVD prevention activities, c) implement a series of evidence-based prevention strategies to be offered in the clinic and community, d) perform both process and outcome evaluations of this demonstration project, and e) compare biologic results (e.g., FRS, lipid levels) with sites not participating in the intervention to assess the effectiveness of our intervention.

ELIGIBILITY:
Inclusion Criteria:

* We will include English or Spanish-speaking individuals between the ages of 30-64 years who actively utilize one of the three community health centers, La Casa Quigg-Newton Family Health Center, the Family and Internal Medicine clinic at the Wellington E. Webb Center for Primary Care, and Westside Neighborhood Health Center for primary care and who have a FRS of 10% or greater. Active utilization will be defined as having 2 or more visits within the past 18 months.

Exclusion Criteria:

* We will exclude pregnant or lactating women, any patient with a prior history of cardiovascular disease (using ICD-9 codes), and/or any patient with a co-morbid illness whose life expectancy less than 12 months (e.g., terminal cancer).

Ages: 30 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 340 (Actual)
Dates: Start 2007-03; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Reduction of CVD risk as measured by Framingham risk score. | within 12-14months after enrollment

SECONDARY OUTCOMES:
Improvement of behavioral and clinical factors that contribute to CVD risk. | 12-14 months after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Judith Shlay, MD, MSPH, Principal Investigator — Denver Health and Hospital Authority; Christopher Urbina, MD, MPH, Principal Investigator — Denver Health and Hospital Authority
Locations (1):
- Denver Health Authority, Denver, Colorado, United States